CLINICAL TRIAL: NCT01260636
Title: A Phase III, Comparative Multi-center Randomized Double-blind, Crossover Study of the Safety, Tolerability and Diagnostic Efficacy of Gadobenate Dimeglumine and Gadopentetate Dimeglumine in Magnetic Resonance Angiography of the Carotid, Renal/Abdominal and Peripheral Arteries
Brief Title: Crossover Comparison of Two Gadolinium Contrast Agents for Use With MRA of Carotid, Renal and Peripheral Arteries
Acronym: VALUE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MH-137
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Carotid, Aortic, Renal or Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — gadobenic acid; Gadolinium DTPA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MultiHance contrast agent (Experimental): MultiHance administered at a dose of 0.1 mmol/kg (0.2 mL/kg)
  Interventions: Drug: Gadobenate Dimeglumine
- Magnevist (Active Comparator): Magnevist administered at a dose of 0.2 mmol/kg
  Interventions: Drug: Gadopentetate Dimeglumine

INTERVENTIONS:
Drug: Gadobenate Dimeglumine — 0.1 mmol/kg, single dose
  Other Names: MultiHance
  Arms: MultiHance contrast agent
Drug: Gadopentetate Dimeglumine — Double dose of 0.2 mmol/kg
  Other Names: Magnevist
  Arms: Magnevist

SUMMARY:
To compare two gadolinium contrast agents in terms of global paired diagnostic preference (primary endpoint) for the assessment of contrast-enhanced MR Angiography of the carotid, renal/abdominal and peripheral arteries

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs of age or older
* referred for enhanced MRA of carotid, renal/abdominal or peripheral arteries
* Able to provide written informed consent and comply with protocol requirements
* Highly suspected of or with known disease of the carotid, renal/abdominal or peripheral vasculature using specific criteria listed in the protocol

Exclusion Criteria:

* pregnant or lactating females
* Known allergy to one or more of the ingredients in the products under investigation
* Significant congestive heart failure ( Class IV)
* Moderate to severe chronic kidney disease
* Therapeutic intervention of any kind for vascular disease in the territory of interest between the two contrast procedures
* Vascular stents in vessels of interest
* Received another contrast agent in the 24 hrs preceding or proceeding each exam
* Previously entered into the study
* Contraindications to MRI
* Severe Claustrophobia Undergone DSA between the two exams

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic Preference | Immediately post dose
  Comparison of a single dose of MultiHance versus the double dose of Magnevist currently used for MR Angiography of the carotid, renal/abdominal/ and peripheral arteries in terms of global diagnostic perference

SECONDARY OUTCOMES:
Safety comparison of two diagnostic agents | UP to 24 hours post dose of each contrast agent
  to compare the safety of the two investigational products in patients undergoing CE-MRA of the carotid, renal/abdominal and peripheral arteries

CONTACTS AND LOCATIONS:
Locations (1):
- Radiology Department Zhongshan Hospital, Fudan University, Shanghai, China

REFERENCES:
- [Derived] Li Y, Li X, Li D, Lu J, Xing X, Yan F, Li Y, Wang X, Iezzi R, De Cobelli F. Multicenter, intraindividual comparison of single-dose gadobenate dimeglumine and double-dose gadopentetate dimeglumine for MR angiography of the supra-aortic arteries (the Supra-Aortic VALUE study). AJNR Am J Neuroradiol. 2013 Apr;34(4):847-54. doi: 10.3174/ajnr.A3298. Epub 2012 Oct 4. PMID 23042922